CLINICAL TRIAL: NCT03834870
Title: Virtual cOaching in Making Informed Choices on Elder Mistreatment Self-Disclosure (VOICES)
Acronym: VOICES
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2000023799; 5R01AG060084-04 (NIH)
Record Dates: First submitted 2018-12-14; First posted 2019-02-08 (Actual); Results first posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-03

CONDITIONS: Elder Abuse
MeSH Terms: interventions — Voice

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elder adults in emergency department setting (Experimental): Elder mistreatment in an Emergency Department setting.
  Interventions: Behavioral: Virtual cOaching in making Informed Choices on Elder Mistreatment Self-Disclosure (VOICES)

INTERVENTIONS:
Behavioral: Virtual cOaching in making Informed Choices on Elder Mistreatment Self-Disclosure (VOICES) — Virtual cOaching in making Informed Choices on Elder Mistreatment Self-Disclosure (VOICES) screening tool.

SUMMARY:
To develop an interactive tool to screen for Elder Mistreatment (EM) in the Emergency Department (ED) to promote self-disclosure.

DETAILED DESCRIPTION:
To develop and refine the interactive VOICES tool, which will promote self-identification and self-disclosure to increase reporting of EM at point-of-care in the Emergency Department (ED) setting. Prior to conducting a feasibility study, focus groups will be conducted to inform the process and to develop a tool to evaluate the use of VOICES.

Feasibility Study: To conduct a feasibility study (N= 800) examining the use of VOICES in a busy ED.

Exploratory Aim: To perform a preliminary evaluation of the accuracy of VOICES as a screening tool in correctly classifying EM cases that were referred to Adult Protective Services (APS).

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older
* Non-full trauma track
* Alert and oriented to person and place
* AMT-4 score of 4
* Able to consent and communicate in English
* Agrees and able to use the iPad
* Not in police custody

Exclusion Criteria:

* subjects who live in nursing homes or other long-term care sitting and do not reside in community setting
* patients will be excluded if they cannot safely undergo the studies required for participation
* subjects with clear signs of EM
* Patient or clinician refusal to participate
* severe hearing and vision impairment
* presenting with active psychotic symptoms
* presenting with acute intoxication
* COVID-19 positive

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1012 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fuad Abujarad, PhD,MSc, Principal Investigator — Yale University
Locations (1):
- St. Raphael Emergency Department, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Elder Adults in Emergency Department Setting
Started | 1012
Completed | 1002
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Elder Adults in Emergency Department Setting
Number analyzed (Participants) | 1002
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.5 (9.04)
Age, Customized [Count of Participants; unit: Participants]
  60-69 | 392
  70-79 | 370
  80-89 | 177
  90+ | 63
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 594
  Male | 408
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 49
  Not Hispanic or Latino | 938
  Unknown or Not Reported | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 298
  White | 673
  More than one race | 16
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 1002
Education [Count of Participants; unit: Participants]
  Associate's Degree | 46
  Undergraduate Degree (Bachelor's program or equivalent) | 192
  Professional Degree (Master's program or equivalent) | 138
  High School Graduate or GED | 290
  High School Not Completed | 92
  Refused/Unknown | 4
  Some college | 240
Household Income [Count of Participants; unit: Participants]
  Less than 25k | 291
  Between 25k to 34k | 122
  Between 35k to 49k | 111
  Between 50k to 74k | 116
  Between 75k to 99k | 63
  Between 100k to 149k | 53
  More than 150k | 42
  Refused/Unknown | 204
Marital Status [Count of Participants; unit: Participants]
  Single or Never Married | 233
  Widowed | 221
  Married or Co-habituating | 360
  Divorced | 157
  Separated | 19
  Other | 7
  Refused/Unknown | 5
Employment Status [Count of Participants; unit: Participants]
  Full Time | 103
  Not Employed/Retired | 840
  Part Time | 56
  Refused/Unknown | 3
Living Arrangement [Count of Participants; unit: Participants]
  In Their Own Home | 936
  In Someone Else's Home | 42
  Assisted Living | 24
Number of Household Members [Median (Standard Deviation); unit: persons] | 2 (1.1)
Internet Usage [Count of Participants; unit: Participants]
  Every Day | 530
  1-2 Times a Week | 157
  1-2 Times a Month | 32
  Rarely | 280
  Refused/Unknown | 3
Confidence in Using Technology [Mean (Standard Deviation); unit: units on a scale] — Confidence in Using Technology is measured by a question that uses a scale of 1-10 (0= Not confident at all, 10= Very confident), where a higher score indicates greater confidence.
  units on a scale | 6.9 (2.91)

OUTCOME MEASURES:

1. Primary Outcome: Implementation in Terms of Participation
Description: Participation will be determined by the ratio of participants who are successfully enrolled to the total number of eligible patients. The numerator, denominator, frequencies and 95% confidence intervals will be reported.
Time Frame: up to 16 months
Population: The total number of eligible participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Elder Adults in Emergency Department Setting
Number analyzed (Participants) | 1204
Participants | 1012
Statistical Analysis 1: Comparison: Elder Adults in Emergency Department Setting; Test type: Other; Percentage of enrolled from eligible = 84.05, 95% CI 2-sided [81.98 to 86.10]

2. Primary Outcome: Implementation in Terms of Usage
Description: Usage will be determined by the number of consented participants enrolled in the study who used VOICES to completion.
Time Frame: up to 16 months
Population: The number of participants who were enrolled in the study (n=1,012)/
Measure: Count of Participants; unit: Participants
Arm/Group | Elder Adults in Emergency Department Setting
Number analyzed (Participants) | 1012
Participants | 1002
Statistical Analysis 1: Comparison: Elder Adults in Emergency Department Setting; Test type: Other; Percentage of enrolled from eligible = 99.01, 95% CI 2-sided [98.40 to 99.60]

3. Other Pre Specified Outcome: Acceptability
Description: Participant satisfaction will be measured along multiple dimensions using post-use satisfaction survey with two 5-point Likert response set scales, developed by the research team.
  Scale 1: Likert scale 1-5, where 1= Very Dissatisfied, and 5= Very Satisfied Scale 2: Likert scale 1-5, where 1= Strongly Disagree, and 5= Strongly Agree
Time Frame: up to 16 months
Population: The number of participants who successfully used VOICES to completion.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Elder Adults in Emergency Department Setting
Number analyzed (Participants) | 1002
units on a scale
  Level of confidentiality and privacy provided while using this tool (Scale 1) | 4.57 (0.76)
  The time it took to complete using the VOICES tool (Scale 1) | 4.44 (0.81)
  Your ability to complete the VOICES tool on your own on the iPad, without any staff (Scale 1) | 4.5 (0.81)
  Time to complete the tool on the iPad was short (Scale 2) | 4.11 (0.98)
  I felt engaged in the tool throughout the process (Scale 2) | 4.29 (0.81)
  Audio and visual aids of the tool were helpful (Scale 2) | 4.41 (0.75)
  I felt the fonts, size and the colors of the text in the tool were appropriate and readable (Scale2) | 4.53 (0.68)
  Using this tool on the iPad was very easy (Scale 2) | 4.53 (0.67)
  I was comfortable answering questions on the iPad (Scale 2) | 4.56 (0.65)
  Using the iPad and the headphones provided more privacy (Scale 2) | 4.5 (0.70)
  I feel comfortable discussing mistreatment with a doctor or medical professional (Scale 2) | 4.4 (0.80)
  This tool is appropriate for learning about mistreatment (Scale 2) | 4.54 (0.66)
  This tool is appropriate to be used in the emergency department (Scale 2) | 4.41 (0.73)
  I was able to complete VOICES on the iPad on my own (Scale 2) | 4.40 (0.80)
  Using VOICES on the iPad was a frustrating experience (Scale 2) | 1.87 (1.30)
  The instructions provided by Vicky were clear and easy to follow (Scale 2) | 4.59 (0.61)
  I feel more confident about understanding EM/resources in case I/someone else I know is mistreated | 4.50 (0.67)
  I feel safer after using VOICES on the iPad (Scale 2) | 4.21 (0.89)
  I learned new, useful things about elder mistreatment (Scale 2) | 4.34 (0.68)
  I would like to see this used by other older adults in the community such as the doctor's office (2) | 4.52 (0.68)

4. Other Pre Specified Outcome: Demand
Description: Demand will be assessed through examining how likely will VOICES be used by patients. To do this, the size of target population of EM victims in the ED will be measured by the % of the patients who self-identified with elder mistreatment and the % who receive the Brief Negotiation Interview (BNI) portion of VOICES.
Time Frame: up to 16 months
Population: The number of participants who successfully used VOICES to completion.
Measure: Count of Participants; unit: Participants
Arm/Group | Elder Adults in Emergency Department Setting
Number analyzed (Participants) | 1002
Participants
  Participants who received the BNI | 71
  Participants who self-identified with elder mistreatment | 67

5. Other Pre Specified Outcome: Practicality
Description: Practicality will be assessed by observing the ease of VOICES use by patients. To do this, a series of steps will be watched to determine the efficiency of implementation measured by the average time (1) to consent & orient participants to the tool and (2) needed to complete VOICES documented by the Research Assistant; and (3) patients perceived time of VOICES as measured on post-survey. Each of these will be reported as part of the overall outcome.
Time Frame: up to 16 months
Population: The number of participants who successfully used VOICES to completion.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Elder Adults in Emergency Department Setting
Number analyzed (Participants) | 1002
minutes
  Actual VOICES Duration | 8.8 (5.4)
  Actual Consent Duration | 14.9 (5.9)
  Participant Estimated Time to Completion | 12.2 (9.1)

6. Other Pre Specified Outcome: Efficacy of the Educational Material
Description: To understand the efficacy of VOICES in this pilot, we will look at how many participants changed their self-identification response after completing the educational component.
Time Frame: up to 16 months
Population: The number of participants who successfully used VOICES to completion.
Measure: Count of Participants; unit: Participants
Arm/Group | Elder Adults in Emergency Department Setting
Number analyzed (Participants) | 1002
Participants
  Overall participants who changed their self-identification response | 40
  "Yes" (does self-identify) response changed to "No" (does not self-identify) response | 21
  "No" (does not self-identify) response changed to "Yes" (does self-identify) response | 19

7. Other Pre Specified Outcome: Efficacy of the Brief Negotiation Interview
Description: We will look at how many patients changed their readiness to disclose after completing the Brief Negotiation Interview (BNI).
Time Frame: up to 16 months
Population: The number of participants who successfully used VOICES to completion and accessed the self-disclosure Brief Negotiation Interview (N=18).
Measure: Count of Participants; unit: Participants
Groups:
- Participants Who Accessed Self-disclosure Brief Negotiation Interview: The group of participants who accessed the customized self-disclosure Brief Negotiation Interview pathway.
Arm/Group | Participants Who Accessed Self-disclosure Brief Negotiation Interview
Number analyzed (Participants) | 18
Participants | 3

8. Other Pre Specified Outcome: Efficacy of Self-Identification on Self-Disclosure
Description: We will explore whether self-identification impacts likelihood of self-disclosure.
  Effect-size estimation measured by change in the % of patients who disclose among those who self-identified.
Time Frame: up to 16 months
Population: The number of participants who self-identified with elder mistreatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Elder Adults in Emergency Department Setting
Number analyzed (Participants) | 67
Participants | 49

9. Other Pre Specified Outcome: Accuracy
Description: To understand the accuracy of the VOICES tool, a preliminary evaluation of the accuracy of VOICES as a screening tool in correctly classifying EM cases that were positive based on social worker assessment, and those referred to Adult Protective Services (APS). The percent correct classification will be reported.
Time Frame: up to 16 months
Population: The number of participants who used VOICES to completion and screened positive for suspicion of elder mistreatment (n=112).
Measure: Count of Participants; unit: Participants
Groups:
- Participant Group Who Screened Positive for Suspicion of Elder Mistreatment: Participant group of overall participants who screened positive for suspicion of elder mistreatment
Arm/Group | Participant Group Who Screened Positive for Suspicion of Elder Mistreatment
Number analyzed (Participants) | 112
Participants
  Participants substantiated for elder mistreatment | 49
  Of the substantiated participants, participants referred to Adult Protective Services (APS): number analyzed (Participants) | 49
  Of the substantiated participants, participants referred to Adult Protective Services (APS) | 11
  Referred APS cases accepted and opened by APS: number analyzed (Participants) | 11
  Referred APS cases accepted and opened by APS | 11

ADVERSE EVENTS:
Time Frame: Up to 16 months
Description: Adverse event data were collected over the entire enrollment period, from 7/20/2020 to 12/01/2021.
Arm/Group | Elder Adults in Emergency Department Setting
All-Cause Mortality (participants affected / at risk) | 0/1012
Serious Adverse Events (participants affected / at risk) | 0/1012
Other Adverse Events (participants affected / at risk) | 0/1012

LIMITATIONS AND CAVEATS:
This study was limited to English-speaking older adults, leading to less representation with the Hispanic/Latino population.

Providers, nurses and other clinical emergency department staff were not included in the study and outcomes only extend to older adult patients in the emergency department.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/70/NCT03834870/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT03834870/SAP_001.pdf
  • Informed Consent Form (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/70/NCT03834870/ICF_002.pdf